CLINICAL TRIAL: NCT04579978
Title: Tumor Immunotherapy and Microbiome Analysis
Acronym: TIME
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Princess Margaret Hospital, Canada (Other); University of Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: TIME
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Advanced Solid Tumor
Keywords: Immune Checkpoint Inhibitor; Microbiome; Immune-Mediated Toxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal samples will be collected for analysis of gut bacteria. Peripheral blood samples will be collected via phlebotomy for analysis of immune markers and circulating bacteria.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with advanced solid tumors starting immunotherapy: Subjects with advanced solid tumors planned to initiate standard of care immune checkpoint inhibitors
- Subjects with advanced solid tumors receiving ICIs: Subjects with advanced solid tumors already receiving standard of care immune checkpoint inhibitors

SUMMARY:
The composition of the gut microbiome has been associated with response and the development of toxicities on immune checkpoint inhibitors (ICIs) in multiple tumor types. The aim of this study is to examine the gut microbiome composition in patients undergoing standard of care treatment for advanced/unresectable and/or metastatic solid tumors with ICIs. Fecal samples and peripheral blood samples will be collected to further characterize the diversity of gut bacteria and to study potential mechanisms by which gut bacteria impact the immune response.

DETAILED DESCRIPTION:
This is a prospective study of gut microbial markers. Patients with histologically confirmed advanced/unresectable or metastatic solid tumors who are planned to initiate standard of care ICIs or are undergoing standard of care treatment with ICIs will be approached for participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Sign written and voluntary informed consent
* Adult patients aged >=18, male or female
* Eastern Cooperative Group (ECOG) performance status 0-2
* Histologic diagnosis of an advanced/unresectable or metastatic solid tumor
* Measurable disease as per RECIST 1.1 criteria
* Be suitable for or receiving ICI treatment
* Prior immunotherapy allowed
* Be willing and able to provide fecal and blood specimens for analysis as per protocol

Exclusion Criteria:

* Subjects with a history of inflammatory bowel disease, chronic diarrhea or malabsorption syndromes and significant prior bowel resection as judged by the study investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with advanced/unresectable or metastatic solid tumors either planned to start standard of care treatment with ICIs or already on treatment with ICIs.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Relative abundance and composition of immunotherapy response-associated bacterial species in patients with advanced/unresectable or metastatic solid tumors | 6 months
  Fecal microbial composition analyzed by 16S rRNA and metagenomic sequencing
Relative abundance and composition of immunotherapy toxicity-associated bacterial species in patients with advanced/unresectable or metastatic solid tumors | 12 months
  Fecal microbial composition analyzed by 16S rRNA and metagenomic sequencing; IgA sequencing of fecal samples from patients who develop diarrhea/colitis

SECONDARY OUTCOMES:
Changes in the composition of the intestinal microbiome induced by ICIs | 6 months
  Fecal microbial composition analyzed by 16S rRNA and metagenomic sequencing
Relative abundance of bacterial DNA in peripheral blood samples | 6 months
  Blood microbial abundance measured via qPCR
Changes in immune cell subsets in the systemic circulation upon progression on ICIs correlated with changes in microbiome composition | 2 years
  Flow cytometry of blood at baseline and at development of progressive disease and analysis of microbiome composition at baseline and at development of progressive disease
Identification of serum metabolites in systemic circulation and correlation with intestinal microbiome composition | 6 months
  Analysis of serum metabolites using chromatography coupled to tandem mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Rossanna C. Pezo, MD/PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No